CLINICAL TRIAL: NCT05666661
Title: Effectiveness of Binaural Beat Technology Combined With Rhythmical Photic Stimulation in Treating Depressive Symptoms in Nurses
Brief Title: Binaural Beat Technology and Rhythmical Photic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Yang Shang-Yu, Assistant professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CMUH110-REC3-021
Record Dates: First submitted 2022-12-09; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Sound; Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sound and light therapy group (BBT and FL group) (Experimental): 30 minutes of intervention every day for 14 consecutive days.
  Interventions: Other: Sound and light therapy (BBT and FL group)
- Sound therapy group (BBT) (Experimental): 30 minutes of intervention every day for 14 consecutive days.
  Interventions: Other: Sound therapy group (BBT)
- Relaxing music group (Sham Comparator): 30 minutes of intervention every day for 14 consecutive days.
  Interventions: Other: Relaxing music group

INTERVENTIONS:
Other: Sound and light therapy (BBT and FL group) — During intervention, the participants close their eyes and wear an eye mask and stereo earphones. They then listen to 30 minutes of 10 Hz BBT music (intercalated with relaxing music) through their mobile phone. The intervention music was first embedded in the participant's mobile phone and the BBT music application was purchased from the mobile phone app (Brainwave Studio software, Dalcoms Inc). When listening to music, 10 Hz light stimulation was added to the BBT and FL group (using a mobile phone). Table 1 shows the intervention status. The rhythmical photic stimulation program was a commercially available mobile phone app (Strobe Therapy software released by FuwhatSoft).
  Arms: Sound and light therapy group (BBT and FL group)
Other: Sound therapy group (BBT) — Participants in the sound therapy group (BBT) listened to 30 minutes of 10 Hz BBT music (intercalated with relaxing music) through their mobile phones. Except for rhythmical photic stimulation, the other steps were the same as the BBT and FL group.
  Arms: Sound therapy group (BBT)
Other: Relaxing music group — Participants listened to 30 minutes of relaxing music (the same as that of the experimental groups) through their mobile phone. Except for rhythmical photic stimulation and 10 Hz BBT, the other steps were the same as the experimental groups.
  Arms: Relaxing music group

SUMMARY:
Background Many nurses must shoulder heavy workloads and often develop depressive emotions due to work stress. Previous studies pointed out that binaural beat technology (BBT) and rhythmical photic stimulation can effectively improve negative emotions but there are very few related empirical studies.

Objectives This study examined the effectiveness of BBT combined with rhythmical photic stimulation in improving depressive symptoms in nurses.

Methods This is a randomized controlled trial and nurses in central Taiwan were recruited as participants. These participants were randomized into three groups: BBT combined with rhythmical photic stimulation group, BBT group, and relaxing music group. The intervention period was 2 weeks, with 30 minutes per session. The Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Index (PSQI), vitality and mental health scale (VT&MH from SF-36), and heart rate variability (HRV) were used as parameters for pre- and posttest evaluation in this study. The Wilcoxon signed-rank test was used to test if there are significant differences in various parameters in the three groups before and after intervention. The Krusal-Wallis test was used to test for significant differences in parameter changes between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* (1) BDI score ≥ 14 points; (2) aged between 20 and 50 years, and (3) did not undergo antidepressant treatment within 3 months before intervention and during intervention.

Exclusion Criteria:

* (1) Subjects with a medical history of mixed psychosis, including schizophrenia, bipolar disorder, and dementia; (2) patients with current acute disease and unstable physiological status; (3) medical history of epilepsy; (4) patients with eye diseases; (5) vertigo (including Meniere's syndrome); (6) hearing loss; and (7) participated in electroconvulsive therapy or transcranial electrical stimulation within 1 month prior to or during intervention.

Ages: 25 Years to 55 Years | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI) | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' homes and the test content was the same as the first test. It took about 10 minutes.
  There were 21 questions in the BDI, and a self-rated method was used for participants to fill in their thoughts in the last 2 weeks. A 4-point Likert scale was used. The score range of each question was 0-3 points. A total score of 0-12 points was normal, 14-19 points was mild depression, 20-28 points was moderate depression, and 29-63 points was severe depression.
Pittsburgh Sleep Quality Index (PSQI) | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' homes and the test content was the same as the first test. It took about 10 minutes.
  There were 18 questions in the PSQI, and participants used a self-rated method to fill in their sleep quality in the last month on a 4-point Likert scale. The total score range was 0-21 points. The higher the score, the poorer the sleep quality. This scale has seven dimensions, including: (1) Subjective sleep quality; (2) Sleep latency; (3) Sleep duration; (4) Sleep efficiency; (5) Sleep disturbances; (6) Daytime dysfunction; and (7) Use of sleep medication. PSQI had good validity and reliability(Tsai et al., 2005).
HRV analyzer | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' homes and the test content was the same as the first test. It took about 5 minutes.
  HRV was used to measure heart rate variability, including five markers: (1) Mean heart rate; (2) SDNN: Standard deviation of all RR intervals, represent the physiological health of autonomic nervous system; the higher the SDNN, the better the physiological health of the autonomic nervous system; (3) nLF: Normalized low frequency, reflects sympathetic nervous activity. The higher the value, the greater the activity; (4) nHF: Normalized high frequency, reflects parasympathetic nervous activity. The higher the value, the greater the activity; (5) LF/HF, a marker reflecting sympathetic and parasympathetic nervous activity.

SECONDARY OUTCOMES:
Vitality scales (VT) | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' homes and the test content was the same as the first test. It took about 10 minutes.
  The vitality (VT) and mental health scales (MH) in SF-36 were used for measurement of secondary outcomes The SF-36 scale covers eight dimensions and 36 questions. Each dimension can be used for testing separately and has good validity and reliability (Yang et al., 2018). The VT and MH scales have four and five questions, respectively. A 6-point Likert scale is used. The score of each question ranges from 1 to 6 points and the total score of the VT and MH scales are 4-24 and 5-30 points, respectively. A higher score indicates better vitality or mental health.
Mental health scales (MH) | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' homes and the test content was the same as the first test. It took about 10 minutes.
  The vitality (VT) and mental health scales (MH) in SF-36 were used for measurement of secondary outcomes The SF-36 scale covers eight dimensions and 36 questions. Each dimension can be used for testing separately and has good validity and reliability (Yang et al., 2018). The VT and MH scales have four and five questions, respectively. A 6-point Likert scale is used. The score of each question ranges from 1 to 6 points and the total score of the VT and MH scales are 4-24 and 5-30 points, respectively. A higher score indicates better vitality or mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Univeraity, Taichung, WuFeng, Taiwan